CLINICAL TRIAL: NCT00588237
Title: A Phase II Study of Intravenous and Intraperitoneal Paclitaxel, Intraperitoneal Cisplatin, and Intravenous Bevacizumab for the Initial Treatment of Optimal Stage II or III Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Brief Title: Intravenous and Intraperitoneal Paclitaxel, Intraperitoneal Cisplatin, and Intravenous Bevacizumab for the Initial Treatment of Optimal Stage II or III Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-064
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Cancer; Primary PERITONEUM; Fallopian Tube Cancer
Keywords: ovary; BEVACIZUMAB; CISPLATIN; TAXOL
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; Cisplatin; Bevacizumab

ARMS (1):
- 1 (Experimental): Paclitaxel, Cisplatin, Bevacizumab
  Interventions: Drug: Paclitaxel,Cisplatin, Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel,Cisplatin, Bevacizumab — IV paclitaxel, followed by IV Bevacizumab on Day 1. Bevacizumab treatment will begin cycle 2, day 1. IP cisplatin will be given on Day 2, and IP Paclitaxel on Day 8. Subjects will receive up to six cycles of therapy, or until disease progression or unacceptable toxicity.

SUMMARY:
The purpose of this study is to test whether it is safe to treat your cancer with 3 drugs instead of 2 drugs. After surgery, your cancer is typically treated with 2 drugs called cisplatin and paclitaxel (also known as Taxol). Cisplatin is given through a port in your belly, and Taxol is given both through the belly port and through the vein (IV). Large clinical studies have shown that this treatment gives the best results for women with your cancer. This treatment, however, also causes many side effects, especially belly pain, nerve injury, lowering of the immune system, and infection risk. In the study you are being asked to join, the dose of Cisplatin will be lower in order to try to lessen these problems. This study will also test the safety of adding a 3rd drug called bevacizumab (also known as Avastin). This drug has been shown to shrink ovarian, peritoneal, or fallopian tube cancer in some patients who have advanced disease, despite having received prior treatment for their cancer. Therefore, it may also be effective in patients, like you, who have a new diagnosis.

Unfortunately, Avastin can cause some dangerous side effects in women with advanced cancer. For instance, it can cause a hole in the intestines, and can increase the risk of blood clots and strokes. Avastin has not been given at the same time as IP therapy, so it is not known if this is a safe or effective combination. In this study, IV Avastin will be given in addition to IP cisplatin, IP Taxol, and IV Taxol, to patients like you who have not had any chemotherapy before. This study aims to find out what effects, good and/or bad, that this combination of drugs has on your body and on your type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed an approved informed consent.
* Subjects with histologic diagnosis of epithelial ovarian carcinoma, primary peritoneal carcinoma, or fallopian tube carcinoma, Stage II or III, with optimal (≤ or equal to 1 cm residual disease) residual disease following initial surgery. All subjects must have had appropriate surgery for ovarian, primary peritoneal, or fallopian tube carcinoma with appropriate tissue available for histologic evaluation to confirm diagnosis and stage. Pathology must be verified at Memorial Sloan-Kettering Cancer Center.
* Subjects with the following histologic epithelial cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma N.O.S.
* Subjects must have a Karnofsky Performance Status (KPS) of ≥ or equal to 70%.
* Subjects must be entered no more than 12 weeks postoperatively.
* Bone marrow function:
* Absolute neutrophil count (ANC) ≥ than or equal to 1,500/µl (equivalent to Common Toxicity Criteria (CTC) Grade 1)
* Platelets ≥ than or equal to 100,000/µl (CTC Grade 0-1)
* Renal function: Creatinine ≤ than or equal to 1.5 mg/dl
* Hepatic function: Bilirubin ≤ than or equal to 1.5 x ULN (CTC Grade 1) AST ≤ than or equal to 2.5 x ULN (CTC Grade 1)
* Neurologic function:Neuropathy (sensory) ≤ than CTC Grade 1
* Urine Protein Creatinine: Urine protein creatinine (UPC) ratio must be < than 1.0 gm. If UPC ratio > than or equal to 1, collection of 24-hour urine measurement of urine protein is recommended as part of the patient's medical management off-study. *
* UPC ratio of spot urine is an estimation of the 24 urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm. UPC ratio is calculated using one of the following formulas:
* [urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/dL
* [(urine protein) x0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L
* The UPCR has been found to correlate directly with the amount of protein excreted in a 24 hour urine collection. Specifically, a UPCR of 1.0 is equivalent to 1.0 gram of protein in a 24 hour urine collection. Obtain at least 4 ml of a random urine sample in a sterile container (does not have to be a 24 hour urine). Send sample to lab with request for urine protein and creatinine levels [separate requests]. The lab will measure protein concentration (mg/dL) and creatinine concentration (mg/dL). The UPCR is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL). Patients must have a UPCR < 1.0 to allow participation in the study.
* Blood coagulation parameters:

PT such that international normalized ratio (INR) is < than or equal to 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a PTT < 1.2 times the upper limit of normal.

* Patients of childbearing potential must have a negative serum pregnancy test prior to study entry and be practicing an effective form of contraception during the study and for at least 6 months after receiving the final treatment of bevacizumab.
* Patients must have an Intraperitoneal (IP) port in place. If a patient does not have an IP port, she must be willing to undergo surgical placement of one.

Exclusion Criteria:

* Subjects with a current diagnosis of epithelial ovarian tumor of low malignant potential (borderline carcinomas) are not eligible. Subjects with a prior diagnosis of a low malignant potential tumor that was surgically resected and who subsequently develop invasive adenocarcinoma are eligible, provided that they have not received prior chemotherapy for any ovarian tumor.
* Subjects who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than 3 years prior to enrollment, and the subject remains free of recurrent or metastatic disease.
* Subjects who have received prior chemotherapy for any abdominal or pelvic tumor are excluded. Subjects may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than 3 years prior to enrollment, and that the subject remains free of recurrent or metastatic disease.
* Patients with synchronous primary endometrial cancer, or a history of primary endometrial cancer, are excluded unless all of the following conditions are met:

  1. Stage not greater than IB.
  2. Less than 3 mm invasion without vascular or lymphatic invasion
  3. No poorly differentiated subtypes, including papillary serous, clear cell or other FIGO grade 3 lesions
* Patients with suboptimal (> 1 cm) residual disease, as determined by the operative surgeon.
* Patients who have received any targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management of their ovarian, peritoneal primary, or fallopian tube cancer.
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, subjects with other invasive malignancies who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy are excluded.
* Subjects with acute hepatitis.
* Subjects with active infection that requires parenteral antibiotics.
* Patients with serious, non-healing wound, ulcer, or bone fracture are not eligible. This includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days. Patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations.
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
* Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months of the first date of treatment on this study.
* Patients with clinically significant cardiovascular disease. This includes:

  1. Uncontrolled hypertension, defined as systolic >150 mm Hg or diastolic > 90 mm Hg
  2. Myocardial infarction or unstable angina < 6 months prior to registration
  3. New York Heart Association (NYHA) Grade II or greater congestive heart failure
  4. Serious cardiac arrhythmia requiring medication
  5. CTCAE grade 2 or greater peripheral vascular disease
* Patients with major surgical procedure, open biopsy, laparoscopy (including intraperitoneal port placement) or significant traumatic injury within 28 days prior to the first date of bevacizumab therapy. Major surgical procedure anticipated during the course of the study. Minor surgical procedures, fine needle aspirates, or core biopsies within 7 days prior to the first date of bevacizumab therapy.
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
* Patients under the age of 18.
* Patients who are pregnant or nursing.
* Evidence of extensive intraperitoneal adhesions at the time of surgery, as determined by the operative surgeon.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Konner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Paclitaxel, Cisplatin, Bevacizumab
Period: Overall Study
Arm/Group | All Patients
Started | 42
Completed | 38
Not Completed | 4
Not completed — Evaluable for toxicity only | 3
Not completed — Patien not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: as determined by the GOG RECIST criteria
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 38
participants
  Complete Response (CR) | 10
  Partial Response (PR) | 13
  Progression Free (P-Free) | 11
  Stable Disease (SD) | 4

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 20/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=42)
ALT, SGPT (Blood and lymphatic system disorders) | 1 (1)
AST, SGOT (Blood and lymphatic system disorders) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Dehydration (General disorders) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Febrile neutropenia (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Necrosis, GI- Small Bowel NOS (Gastrointestinal disorders) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1)
Obstruction, GI- Small bowel NOS (Gastrointestinal disorders) | 4 (4)
Pain - Abdomen NOS (General disorders) | 2 (2)
Pain - Back (General disorders) | 1 (1)
Pain - Head/headache (General disorders) | 1 (1)
Perforation, GI- Colon (Gastrointestinal disorders) | 1 (1)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vasovagal episode (Nervous system disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wound complication, non-infectious (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=42)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (5)
ALT, SGPT (Metabolism and nutrition disorders) | 6 (6)
AST, SGOT (Metabolism and nutrition disorders) | 3 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 13 (13)
Creatinine (Metabolism and nutrition disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 30 (30)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 33 (33)
Hemoglobin (Blood and lymphatic system disorders) | 27 (27)
Hypertension (Cardiac disorders) | 10 (10)
Hypotension (Cardiac disorders) | 4 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 20 (20)
Lymphopenia (Blood and lymphatic system disorders) | 10 (10)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 9 (9)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 15 (15)
Neuropathy: sensory (Nervous system disorders) | 8 (8)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 24 (24)
Obstruction, GI- Small bowel NOS (Gastrointestinal disorders) | 4 (4)
Pain - Abdomen NOS (General disorders) | 13 (13)
Pain - Back (General disorders) | 3 (3)
Pain - Head/headache (General disorders) | 4 (4)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 10 (10)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 4 (4)
Platelets (Blood and lymphatic system disorders) | 3 (3)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (5)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 4 (4)
Prothrombin time international normalized ratio (INR) (Blood and lymphatic system disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 4 (4)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 6 (6)
Tinnitus (Ear and labyrinth disorders) | 6 (6)
Vasovagal episode (Nervous system disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 11 (11)
Weight gain (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes